CLINICAL TRIAL: NCT03693963
Title: PRospective Study for the TrEatment of Atherosclerotic Lesions in the Infrapopliteal Arteries Using the Serranator® DevicE: PRELUDE BTK (Below The Knee) Study
Brief Title: The PRELUDE BTK Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cagent Vascular LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-0197
Record Dates: First submitted 2018-07-20; First posted 2018-10-03 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2020-01

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single Arm, treated with Serranator (Other): Subjects treated with Serrantor
  Interventions: Device: Serranator

INTERVENTIONS:
Device: Serranator — The Serranator® PTA Serration Balloon Catheter is an over-the-wire (OTW) balloon dilatation catheter designed to perform percutaneous transluminal angioplasty (PTA) for peripheral indications.

SUMMARY:
The objective of the PRELUDE BTK study is to assess safety and efficacy of the Serranator® PTA Serration Balloon Catheter (study device) in subjects with atherosclerotic peripheral artery disease of the infrapopliteal arteries.

DETAILED DESCRIPTION:
Single arm, prospective, multi-center feasibility study enrolling up to 48 subjects with atherosclerotic lesions in the infrapopliteal arteries and/or Critical Limb Ischemia (CLI). The study will capture acute angiographic data to compare the pre-Serranator® inflation vs post inflation effects and will include 6 month clinical follow up.

The study population will consist of subjects with claudication or CLI, with de novo stenoses or non-stented restenotic or total occlusion lesions in infrapopliteal arteries having lesion length up to and including 12 cm in length and reference vessel diameter of 2.5 mm to 3.5 mm inclusive.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of >18 years old.
2. Women of child bearing potential must have a negative urine pregnancy test within 7 days of index procedure.
3. Subject or subject's legal representative has been informed of the nature of the study, agrees to participate and comply with all follow-up visits and has signed the consent form.
4. Subject is eligible for standard surgical repair in target limb if necessary.
5. Subject has Rutherford Clinical Category 3, 4 or 5. Enrollment of Rutherford 3 will be limited to no more than 40% of total subjects.
6. Estimated life expectancy > 1 year.

Angiographic Inclusion Criteria:

1. Target lesion(s) has stenosis >70% by visual assessment;
2. De-novo, or non-stented re-stenotic lesions;
3. Reference vessel diameter is between 2.5 mm and 3.5 mm, inclusive;
4. Target lesions involve infra-popliteal tibial arteries above the tibio-talar joint;
5. Up to two target lesion(s) may be treated. These target lesions may be located in a single or two infrapopliteal arteries;
6. A target lesion may consist of one long or multiple serial lesions that are up to and including 12 cm in length that can be covered by a single balloon (longest balloon length for this study will be 12 cm);
7. If more than one critical lesion is identified in two different vessels but only one lesion matches the inclusion criteria, that lesion should be treated as the target lesion and the other non-qualifying lesion in the other vessel may be treated with commercial devices in any manner the investigator decides except by atherectomy;
8. If two critical lesions are identified in two vessels and both qualify for the study, the investigator may treat both lesions with investigational balloons or may choose to identify one lesion as the target lesion and treat the second lesion with commercial devices except atherectomy;
9. If two critical lesions are in one vessel and both lesions qualify for the study, both lesions should be treated with investigational balloons. Lesions that are within 3 cm of each other will be treated as a single lesion;
10. Target vessel(s) reconstituted at or above the ankle with inline flow to at least one patent inframalleolar outflow vessel in each target vessel. If the peroneal artery is the treated artery, it should supply collaterals at the ankle that reconstitute an inframalleolar outflow vessel;
11. Successful treatment of inflow stenosis (DS>50%), from the iliac to the target lesion. Stenosis can be treated during the same procedure using standard angioplasty, DCB, DES, and/or stenting but use of atherectomy is excluded. The inflow lesion(s) must be treated first, prior to consideration of treatment of the target lesion. Subject can be enrolled if the inflow lesion(s) are treated and results in <30% residual stenosis and no evidence of embolization or significant complications.

Exclusion Criteria:

1. Rutherford Clinical Category 1, 2, or 6
2. Evidence of aneurysm or acute thrombus in the target vessel.
3. Subjects with previous bypass surgery in lower target extremity.
4. Planned major amputation (above the ankle) of either limb.
5. Subject has significant stenosis or occlusion of inflow tract not successfully treated (>30% residual stenosis and/or significant complication of the procedure).
6. History of any open surgical procedure within the past 30 days.
7. Planned endovascular procedure within 14 days prior to the BTK procedure, except to treat the inflow vessels on the day of the procedure, or a planned endovascular or open surgical procedure within the next 30 days after the BTK procedure on either limb.
8. Planned intervention of occluded or stenotic pedal arteries at the time of the index procedure.
9. Subject has an allergy to contrast medium that cannot be pretreated.
10. Episode of acute limb ischemia within past 30 days.
11. Subject has systemic infection with positive blood cultures/ bacteremia within one week.
12. Subject has a hypercoagulable disorder
13. Subject in whom antiplatelet, anticoagulant, or thrombolytic therapy is contraindicated.
14. Myocardial infarction within 30 days prior to enrollment.
15. History of stroke or TIA within 90 days prior to enrollment.
16. Subject has acute or chronic renal disease (e.g., as measured by a serum creatinine of >2.5 mg/dL or >220 umol/L).
17. Subject is pregnant or breastfeeding.
18. Subject is participating in another research study of a device, medication, which could, in the opinion of the investigator, affect the results of this study.
19. Subject has other medical, social or psychological problems that in the opinion of the investigator would preclude them from receiving this treatment and the procedures and or participating in evaluations pre- and post-treatment.
20. Thrombolysis of the target vessel within 72 hours prior to the index procedure, where complete resolution of the thrombus was not achieved.
21. Known allergies to both antiplatelet agents, aspirin, or heparin.
22. History of neutropenia, coagulopathy, or thrombocytopenia that was unexplained or is considered to be at risk for reoccurrence.
23. Platelet count less than 80,000/μL.
24. Subject requires general anesthesia for the procedure.
25. Subject requires dialysis.
26. Subject has heel gangrene and anything worse than WIfI 2.

Angiographic Exclusion Criteria:

1. De-novo, or non-stented re-stenotic lesions or Chronic Total Occlusions (CTO) > 12 cm in length.
2. Acute Total Occlusions; evidence of acute thrombus formation by angiography.
3. In-stent restenotic lesions.
4. Inability to cross the lesion with a guidewire.
5. Atherectomy for inflow treatment or planned use in below the knee vessel(s)
6. Intended use of adjunctive primary treatment modalities of target lesion(s) (atherectomy, laser, cutting balloons, DCBs, stents).
7. If two critical lesions are in one vessel but only one lesion qualifies, and the other does not, the subject should not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-04-11 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Incidence of MALE and POD (Safety) | 30 days post procedure
  Composite of Major Adverse Limb Events (MALE) and Peri-procedural Death (POD), assessed at 30 days post procedure. MALE plus POD is defined as a composite of all cause death, thrombolysis/thrombectomy at the target lesion, open surgical revision or bypass, and major (above ankle) target limb amputation at 30 days post procedure. Safety will be evaluated on a per subject basis.

SECONDARY OUTCOMES:
Rate of Device Success (Procedural Efficacy) | Immediately Post Serranator treatment
  Procedural efficacy will be assessed by the rate of device success defined as the achievement of successful insertion, balloon inflation and deflation, and removal of the study device(s) with a final diameter stenosis of <50% by visual assessment at the intended target site using only the Serranator device. Device success will be evaluated on a per lesion basis.

CONTACTS AND LOCATIONS:
Locations (6):
- Medical University of Graz, Graz, Austria
- Germany (3):
  - Klinikum Hochsauerland GmbH, Arnsberg
  - Krankenhaus Buchholz, Buchholz
  - Imland Klinik Rendsburg, Rendsburg
- Auckland City Hospital, Auckland, Grafton, New Zealand
- Polsko-Amerykańskie Kliniki Serca PAKS, Chrzanów, Poland

IPD SHARING:
Plan to Share IPD: No